CLINICAL TRIAL: NCT04546321
Title: Comparative Study Between Serum Level of Total L Carnitine in Neonatal Hypoxic Ischemic Encephalopathy (HIE) and Transient Tachypnea of the Newborn (TTN)
Brief Title: Measuring Serum Level of Total L Carnitine in HIE and TTN
Acronym: HIELcarnitine
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amira Shalaby, Lecturer of Pediatrics and Neonataology, Assiut University
Other Study IDs: Assiut U CH
Record Dates: First submitted 2020-09-05; First posted 2020-09-14 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: Compare Between the Serum Level of Lcarnitine in HIE Cases and TTN
Keywords: HIE,Lcarnitine level,TTN

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 1 ml of newborn serum frozen to be analyzed by human ELIZA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HIE group (I): All fullterm newborn admitted to the NICU with Hypoxic Ischemic Encephalopathy during the study period
  Interventions: Other: serum L carnitine level measuring
- TTN group(II): All fullterm babies with Transient Tachypnea of the Newborn admitted to the NICU during the study period
  Interventions: Other: serum L carnitine level measuring

INTERVENTIONS:
Other: serum L carnitine level measuring — The serum level of total L carnitine was measured for both HIE and TTN cases

SUMMARY:
It is a comparative prospective and observational study conducted at Neonatal Intensive Care Unit (NICU) in Assiut University Children Hospital. All cases of perinatal asphyxia and TTN admitted to the NICU during the period 12-2016 to 6-2018 were included. All the included newborns were examined and the serum level of total L carnitine was measured. Then we compared the demographic data and investigation of cases with HIE with the outcome of those cases. Results: It was found that serum level of total L carnitine decreased in both HIE and TTN cases but without significant difference with mean 5.51 ± 1.30 umol/l in group I vs 6.22 ± 2.56 umol/l in group II. The male factor with changes in the serum sodium (132.63 ± 9.30) and abnormal serum creatinine level [1.4 (0.7-15.0)] were significantly related to the outcome of cases with HIE

DETAILED DESCRIPTION:
This is a prospective comparative and observational study included all the full-term HIE and TTN cases admitted to NICU of the University Children Hospital during the period of December 2016 to June 2018. The newborns with perinatal asphyxia who died before admission, gestational age<37wks and those with congenital anomalies were excluded. The study included 35 HIE Patients and 12 TTN patients. All cases were subjected to full perinatal history and clinical examination. HIE cases were classified clinically by Sarnat staging (Sarnat and Sarnat, 1976) [10]. HIE cases were subjected to investigations as capillary blood gases, complete blood count (CBC), and electrolytes, renal function. The demographic data and the results of HIE investigations will be correlated to the outcome. The serum level of total L carnitine was measured for both HIE and TTN cases by sending 1 ml of newborn serum frozen to be analyzed by human ELIZA (Enzyme Linked Immunosorbent Assay) kit (SinoGeneClon Biotech Co.,Ltd) within the 1st week of life and compared with each other. Normal range in males and females 17.4-58.7umol/l. the

Statistical analysis:

Data entry and data analysis were done using SPSS version 22 (Statistical Package for Social Science). Data were presented as number, percentage, mean, standard deviation and median. Chi-square and Fisher Exact tests were used to compare between qualitative variables. Independent samples t-test was used to compare quantitative variables between two groups and ANOVA test for more than two groups in case of parametric data. Mann-Whitney test was used to compare quantitative variables between groups in case of non-parametric data. P-value considered statistically significant when P < 0.05.

Results:

The study included 35 cases of HIE (group I) and 12 cases of TTN (group II) all cases were full-term babies there was no significance between the two groups in the demographic data (sex, weight and maternal age) . There were (19) 54.3% females and (16) 47.7% males in the first group versus 33.3% females and 66.7% males in the 2nd group.The mean birth weight for the first group was 2.78 ± 0.50 kg versus 2.86 ± 0.28 kg in the second group. There were 22 cases and 11 cases delivered by cesarean section in the 1st group and the 2nd group respectively. There were 13 cases and 1 case delivered by normal vaginal delivery in group I and group II respectively. On comparison between the two groups in measuring the serum level of total L carnitine. The serum level of total L carnitine had decreased in both groups with a mean of 5.51 ± 1.30 umol/l in group I versus 6.22 ± 2.56 umol/l in group II. Then after correlation between the demographic data and investigations of cases of HIE with the outcome there was a significant correlation between male factor and death by deaths of 66% of males with HIE and also there was a significant correlation between the outcome and grade III of HIE ( 86.7% of grade III died) .There were a significant correlation between hyponatremia (132.63 ± 9.30) with death of HIE cases and abnormal serum creatinine [1.4 (0.7-15.0)] with death of HIE cases.

ELIGIBILITY:
Inclusion Criteria:

* all the full-term HIE and TTN cases admitted to NICU of the University Children Hospital during the period of December 2016 to June 2018.

Exclusion Criteria:

* The newborns with perinatal asphyxia who died before admission, gestational age<37wks and those with congenital anomalies were excluded

Ages: 1 Minute to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: fulllterm newborn admitted to the NICU
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
comparison | 18 months
  The serum level of total L carnitine was measured for both HIE and TTN cases

SECONDARY OUTCOMES:
correlation | 7-10 days
  . The demographic data and the results of HIE investigations will be correlated to the outcome

CONTACTS AND LOCATIONS:
Overall Officials: Amira Shalaby, Principal Investigator — NICU,Assiut University Children Hospital

IPD SHARING:
Plan to Share IPD: Yes
To share the IPD related to the results
Supporting Information: CSR
Time Frame: after publication